CLINICAL TRIAL: NCT00222001
Title: Outcome Evaluation of Triage for Health Maintenance Organization (HMO) Patients Performed by Doctors in a Medical Telemedicine Center
Brief Title: Telephone Triage Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Medgate AG, Switzerland (Unknown); HMO Gesundheitsplan Basel, Switzerland (Unknown)
Responsible Party: Sponsor
Other Study IDs: MS-001-2002
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Any Medical Condition Presented by Patient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HMO Patients: Measurement of telephone triage outcome.

SUMMARY:
The advance of communication technology has changed medical practice. The concept of medical telemedicine centers receiving, assessing and managing calls from patients or their carers on a 24 hour, 7 days a week basis is spreading in the US as well as in European countries. Usually specially trained nurses using dedicated decision support software provide the service. One aspect is the so-called triage, i.e. the decision on urgency and optimal treatment path of a stated medical problem, which has the potential to contain overall treatment costs.

Despite proliferation of these services, little is known about the quality of the services provided.

In October 2000 the first 24-hour medical telemedicine centre staffed by medical doctors started operating in Switzerland. The aims of this study are to assess the quality of service provided by doctors using decision support software and to determine potential predictors of incorrect triage.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Insured with HMO Basel
* Patient of HMO practise Sternengasse
* First call to Medgate for a given medical problem
* Call is a telephone triage
* Informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Regular HMO patients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2002-12; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Correctness of triage decision | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Serge O Reichlin, MD, Principal Investigator — University Hospital Basel and Medgate AG
Locations (2):
- Switzerland (2):
  - Medgate, Basel, Basel
  - University Hospital Basel, Basel